CLINICAL TRIAL: NCT04120623
Title: Therapeutic Effect of Dapagliflozin Combined With CSII on Newly Diagnosed Type 2 Diabetes Mellitus With Continuous Glucose Monitoring System
Brief Title: Therapeutic Effect of Dapagliflozin Combined With CSII on Newly Diagnosed Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20190926-03
Record Dates: First submitted 2019-09-29; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Continuous Glucose Monitoring System (CGMS); Dapagliflozin; Continuous Subcutaneous Insulin Infusion ( CSII)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin combined with CSII (Experimental): Dapagliflozin 10MG combined with Aspart infused by CSII as glucose lowering therapy.
  Interventions: Drug: Dapagliflozin 10 MG
- CSII alone (Active Comparator): Aspart infused by CSII alone as glucose lowering therapy.
  Interventions: Drug: Insulin Aspart

INTERVENTIONS:
Drug: Dapagliflozin 10 MG — Dapagliflozin 10 MG combined with Insulin Aspart infused by continuous subcutaneous insulin infusion ( CSII).
  Other Names: Dapagliflozin combined with CSII
  Arms: Dapagliflozin combined with CSII
Drug: Insulin Aspart — Insulin Aspart is infused through continuous subcutaneous insulin infusion ( CSII)
  Other Names: CSII alone
  Arms: CSII alone

SUMMARY:
To compare the effect of dapagliflozin combined with CSII and CSII alone on glucose profile in newly diagnosed type 2 diabetes mellitus by continuous glucose monitoring system.

DETAILED DESCRIPTION:
To compare the effect of dapagliflozin combined with continuous subcutaneous insulin infusion (CSII) and CSII alone on glucose profile in newly diagnosed type 2 diabetes mellitus by continuous glucose monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* volunteer to participate and be able to sign informed consent prior to the trial.
* patients with type 2 diabetes or type 1 diabetes, aged 18-80 years old.
* No acute complications such as diabetic ketoacidosis, diabetic hyperosmolar syndrome, etc.
* Subjects are able and willing to monitor peripheral blood sugar and regularity of diet and exercise.

Exclusion Criteria:

* Patients with insulin allergy.
* Impaired liver and kidney function with ALT 2.5 times higher than the upper limit of normal value; Serum creatinine was 1.3 times higher than the upper limit of normal.
* Drug abuse and alcohol dependence in the past 5 years.
* Systemic hormone therapy was used in the last three months.
* Patients with poor compliance and irregular diet and exercise.
* Patients with pregnancy, lactation or pregnancy intention.
* Any other obvious conditions or associated diseases determined by the researcher: such as severe cardiopulmonary diseases, endocrine diseases, neurological diseases, tumors and other diseases, other pancreatic diseases, history of mental diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
the effect of dapagliflozin combined with CSII on glucose profile | 5 weeks
  To compare the effect of dapagliflozin combined with CSII and CSII alone on glucose profile(the mean amplitude of glycemic excursions(MAGE),The 24-hrs mean glucose(MG) ) in newly diagnosed type 2 diabetes mellitus by continuous glucose monitoring system

SECONDARY OUTCOMES:
the effects of dapagliflozin combined with CSII on weight | 5 weeks
  To compare the effect of dapagliflozin combined with CSII and CSII alone on weight in kilogram
the effects of dapagliflozin combined with CSII on blood pressure | 5 weeks
  To compare the effect of dapagliflozin combined with CSII and CSII alone on blood pressure in mmHg
the effects of dapagliflozin combined with CSII on lipid metabolism(total cholesterol in mmol/l, total glyceride in mmol/l) | 5 weeks
  To compare the effect of dapagliflozin combined with CSII and CSII alone on lipid metabolism(total cholesterol in mmol/l, total glyceride in mmol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Ma, Study Director — Nanjing First Hospital, Affiliated to Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No